CLINICAL TRIAL: NCT04579523
Title: A Phase I Trial Evaluating Escalating Doses of ²¹¹At-Labeled Anti-CD38 Monoclonal Antibody Followed by HLA-Matched or Haploidentical Donor Hematopoietic Cell Transplantation for High-Risk Multiple Myeloma
Brief Title: ²¹¹At-OKT10-B10 and Fludarabine Alone or in Combination With Cyclophosphamide and Low-Dose TBI Before Donor Stem Cell Transplant for the Treatment of Newly Diagnosed, Recurrent, or Refractory High-Risk Multiple Myeloma
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG1121028; NCI-2020-06835 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10467 (Other: Fred Hutch/University of Washington Cancer Consortium); P01CA078902 (NIH)
Record Dates: First submitted 2020-09-23; First posted 2020-10-08 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-06

CONDITIONS: Multiple Myeloma; Recurrent Multiple Myeloma; Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Stem Cell Transplantation; Cyclophosphamide; fludarabine phosphate; Whole-Body Irradiation; X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (²¹¹At-OKT10-B10, fludarabine, TBI, HCT) (Experimental): Patients with HLA-matched related or unrelated donors receive ²¹¹At-OKT10-B10 IV on day -7 (day -10 to -5) and fludarabine IV over 30 minutes on days -4 to -2. Patients then undergo TBI and allogeneic HCT on day 0.
  Additionally, patients undergo x-rays on study, and blood sample collection, bone marrow biopsy, and bone marrow aspiration throughout the study.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Biological: Astatine At 211 Anti-CD38 Monoclonal Antibody OKT10-B10; Drug: Fludarabine Phosphate; Radiation: Total-Body Irradiation; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: X-Ray Imaging
- Arm B (²¹¹At-OKT10-B10, chemotherapy, TBI, HCT) (Experimental): Patients with HLA-matched haploidentical donors receive ²¹¹At-OKT10-B10 IV on day -8 (day -14 to -7), fludarabine IV over 30 minutes on days -6 to -2, and cyclophosphamide IV over 1 hour on day -6 and -5. Patients then undergo TBI on day -1 and allogeneic HCT on day 0.
  Additionally, patients undergo x-rays on study, and blood sample collection, bone marrow biopsy, and bone marrow aspiration throughout the study.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Biological: Astatine At 211 Anti-CD38 Monoclonal Antibody OKT10-B10; Drug: Cyclophosphamide; Drug: Fludarabine Phosphate; Radiation: Total-Body Irradiation; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: X-Ray Imaging

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo HCT
  Other Names: Allogeneic; Allogeneic Hematopoietic Cell Transplantation; Allogeneic Stem Cell Transplantation; HSC; HSCT; Stem Cell Transplantation, Allogeneic
Biological: Astatine At 211 Anti-CD38 Monoclonal Antibody OKT10-B10 — Given IV
  Other Names: ²¹¹At-OKT10-B10; [²¹¹At]OKT10-B10; Astatine 211-labeled Anti-CD38 Monoclonal Antibody OKT10-B10; Astatine At 211 Anti-CD38 MoAb OKT10-B10; Astatine-211-OKT10-B10; At211-OKT10-B10
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
  Arms: Arm B (²¹¹At-OKT10-B10, chemotherapy, TBI, HCT)
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: SCT_TBI; TBI; Total Body Irradiation; Whole Body Irradiation; Whole-Body Irradiation
Procedure: Biospecimen Collection — Undergo blood collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspirate
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
Procedure: X-Ray Imaging — Undergo chest x-rays
  Other Names: X-RAY

SUMMARY:
This phase I trial investigates the side effects and best dose of ²¹¹At-OKT10-B10 when given together with fludarabine, alone or in combination with cyclophosphamide and low-dose total-body irradiation (TBI) before donor stem cell transplant in treating patients with high-risk multiple myeloma that is newly diagnosed, has come back (recurrent), or does not respond to treatment (refractory). ²¹¹At-OKT10-B10 is a monoclonal antibody, called OKT10-B10, linked to a radioactive agent called ²¹¹At. OKT10-B10 attaches to CD38 positive cancer cells in a targeted way and delivers ²¹¹At to kill them. Chemotherapy drugs, such as fludarabine and cyclophosphamide, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy such as TBI uses high energy x-rays to kill cancer cells and shrink tumors. Giving ²¹¹At-OKT10-B10 together with chemotherapy and TBI before a donor stem cell transplant helps kill cancer cells in the body and helps make room in the patient's bone marrow for new blood-forming cells. When the healthy stem cells from a donor are infused into a patient, they may help the patient's bone marrow make more healthy cells and platelets and may help destroy any remaining cancer cells.

DETAILED DESCRIPTION:
OUTLINE: This is a dose-escalation study of ²¹¹At-OKT10-B10. Patients are assigned to 1 of 2 arms.

ARM A: Patients with HLA-matched related or unrelated donors receive ²¹¹At-OKT10-B10 intravenously (IV) on day -7 (day -10 to -5) and fludarabine IV over 30 minutes on days -4 to -2. Patients then undergo TBI and allogeneic HCT on day 0. Additionally, patients undergo x-rays on study, and blood sample collection, bone marrow biopsy, and bone marrow aspiration throughout the study.

ARM B: Patients with HLA-matched haploidentical donors receive ²¹¹At-OKT10-B10 IV on day -8 (day -14 to -7), fludarabine IV over 30 minutes on days -6 to -2, and cyclophosphamide IV over 1 hour on day -6 and -5. Patients then undergo TBI on day -1 and allogeneic HCT on day 0. Additionally, patients undergo x-rays on study, and blood sample collection, bone marrow biopsy, and bone marrow aspiration throughout the study.

After completion of study treatment, patients are followed up at 9, 12, 18 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed or relapsed/refractory multiple myeloma
* Patients with multiple myeloma must have at least one of the following high-risk features:

  * t(4;14), t(14;16), t(14;20) or deletion 17p, gain in chromosome 1q (> 3 copies of CKS1b) by fluorescence in situ hybridization (FISH); hypodiploidy; complex karyotype
  * Revised International Staging System III
  * Plasmablastic morphology
  * History of primary or secondary plasma cell leukemia
* Patients must start ²¹¹At-OKT10-B10 within 40-180 days of autologous stem cell transplant (either as part of their induction, or as salvage)
* Patients must have an estimated creatinine clearance greater than 50/ml per minute measured by 24-hour urine collection
* Total bilirubin < 2 times the upper limit of normal
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2 times the upper limit of normal)
* Patients must have an Eastern Cooperative Oncology Group (ECOG) =< 2 or Karnofsky >= 70
* Patients must have CD38+ myeloma cells as demonstrated by either flow cytometry or immunohistochemistry in most recent bone marrow that had evidence of clonal plasma cells
* For patients of childbearing potential, must have a negative urinary pregnancy test on the day of and prior to infusion of ²¹¹At-OKT10-B10
* Ability to provide informed consent
* Patients must have an HLA-matched related donor or an HLA-matched unrelated donor who meets standard Fred Hutchinson Cancer Center and/or National Marrow Donor Program (NMDP) or other donor center criteria for peripheral blood stem cell (PBSC) or bone marrow donation, as follows:

  * Related donor: related to the patient and genotypically or phenotypically identical for HLA-A, B, C, DRB1 and DQB1. Phenotypic identity must be confirmed by high-resolution typing
  * Unrelated donor:

    * Matched for HLA-A, B, C, DRB1 and DQB1 by high resolution typing; OR
    * Mismatched for a single allele without antigen mismatching at HLA-A, B, or C as defined by high resolution typing but otherwise matched for HLA-A, B, C, DRB1 and DQB1 by high resolution typing
    * Donors are excluded when preexisting immunoreactivity is identified that would jeopardize donor hematopoietic cell engraftment. The recommended procedure for patients with 10 of 10 HLA allele level (phenotypic) match is to obtain panel reactive antibody (PRA) screens to class I and class II antigens for all patients before HCT. If the PRA shows > 10% activity, then flow cytometric or B and T cell cytotoxic cross matches should be obtained. The donor should be excluded if any of the cytotoxic cross match assays are positive. For those patients with an HLA class I allele mismatch, flow cytometric or B and T cell cytotoxic cross matches should be obtained regardless of the PRA results. A positive anti-donor cytotoxic crossmatch is an absolute donor exclusion
    * Patient and donor pairs homozygous at a mismatched allele in the graft rejection vector are considered a two-allele mismatch, i.e., the patient is A*0101 and the donor is A*0102, and this type of mismatch is not allowed
* Patients without an HLA-matched related or unrelated donor available must have a related donor who is identical for one HLA haplotype and mismatched at the HLA-A, -B or DRB1 loci of the unshared haplotype with the exception of single HLA-A, -B or DRB1 mismatches

Exclusion Criteria:

* History of central nervous system involvement by multiple myeloma
* Presence of circulating plasma cells in the peripheral blood of 5% or more by flow cytometry or morphology
* Prior radioimmunotherapy or radiation of > 20 Gy to pelvis or at maximally tolerated levels to any critical normal organ
* Prior allogeneic HCT
* More than two prior autologous HCTs
* Patients with plasmacytomas > 1 cm in bone marrow or any extramedullary plasmacytoma. Previously fludeoxyglucose F-18 (FDG) avid mass lesions by positron emission tomography (PET) that are no longer hypermetabolic following the most recent cycle of therapy are exempt, as are plasmacytomas irradiated with curative intent (>= 35 Gy)
* Patients with symptomatic coronary artery disease defined as having angina or anginal equivalent, and/or arrhythmias requiring anti-arrhythmics for rhythm control
* History of reactive airway disease and clinically significant asthma requiring ongoing treatment
* Patients with the following organ dysfunction:

  * Left ventricular ejection fraction < 40% in patients with HLA-matched or unrelated donor or < 45% in patients with an HLA-haploidentical donor
  * New York Heart Association (NYHA) class > 1 heart failure
  * Corrected diffusing capacity of the lungs for carbon monoxide (DLCO) < 50% or receiving supplemental continuous oxygen. When pulmonary function tests cannot be obtained, the 6-minute walk test (6MWT, also known as exercise oximetry) will be used: Any patient with oxygen saturation on room air of < 90% during a 6MWT will be excluded
  * Liver abnormalities: fulminant liver failure, cirrhosis of the liver with evidence of portal hypertension, alcoholic hepatitis, esophageal varices, hepatic encephalopathy, uncorrectable hepatic synthetic dysfunction as evidenced by prolongation of the prothrombin time, ascites related to portal hypertension, bacterial or fungal liver abscess, biliary obstruction, chronic viral hepatitis, or symptomatic biliary disease
* Patients who are known to be seropositive for human immunodeficiency virus (HIV)
* Perceived inability to tolerate diagnostic or therapeutic procedures
* Women of childbearing potential who are pregnant (beta-human chorionic gonadotropin [HCG]+) or breast feeding
* Fertile men and women unwilling to use contraceptives during and for 12 months post-transplant
* Uncontrolled or untreated active infection
* Patients with known AL subtype amyloidosis
* Inability to understand or give an informed consent
* Known allergy to murine-based monoclonal antibodies
* Known contraindications to radiotherapy
* History of another primary malignancy that has not been in remission for at least 2 years. The following are exempt from the 2-year-limit: nonmelanoma skin cancer, curatively treated localized prostate cancer, or cervical carcinoma in situ or squamous intraepithelial lesion on papanicolaou (PAP) smear
* Therapy with anti-CD38 monoclonal antibody within 3 months of ²¹¹At-OKT10-B10 infusion
* Prior therapy with radiolabeled monoclonal antibodies
* Any history of treatment with checkpoint inhibitor/s

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of radiation delivered via ²¹¹At-OKT10-B10 | Up to 100 days following HCT
  MTD is defined as the dose of ²¹¹At-OKT10-B10 associated with a true dose limiting toxicity (DLT) rate of 25%, where DLT is defined as grade III/IV regimen-related toxicity according to the Bearman Scale.

SECONDARY OUTCOMES:
Disease response | Between days 70 to 90 post-transplant
  Definition of disease status will be performed using the established International Myeloma Working Group (IMWG) response criteria for stringent complete response, complete response, partial response (PR) and no response. Relapse is defined per IMWG criteria. The response rates (PR or better) will be estimated along with the exact 95% confidence interval.
Duration of response | From date of response assessment (days +70-90 following allogeneic HCT) until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  Duration of response will be estimated using Kaplan-Meier methodology.
Minimal residual disease (MRD) | Between days 70 to 90 post-transplant
  MRD will be assessed in the comprehensive response evaluation/restaging. The proportion who achieve MRD will be estimated along with an exact 95% confidence interval.
One-year disease -free survival | From allogeneic hematopoietic cell transplantation to disease progression, relapse or death, assessed at 1 year
  Kaplan-Meier methodology will be used to estimate the 1-year disease-free survival.
One-year overall survival (OS) | From transplantation to death or last patient contact, assessed at 1 year
  Kaplan-Meier methodology will be used to estimate the 1-year OS.

CONTACTS AND LOCATIONS:
Overall Officials: Phuong Vo, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No